CLINICAL TRIAL: NCT01130649
Title: Pilot Study of Real-time Automated Tracking System for Patients With Epilepsy
Brief Title: Remote Tracking of Epilepsy Patients
Status: Withdrawn | Type: Observational
Why Stopped: not funded
Sponsor: University of California, San Francisco (Other)
Collaborators: San Francisco Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, John Hixson, Associate Professor of Neurology, University of California, San Francisco
Other Study IDs: Epitrack
Record Dates: First submitted 2010-05-24; First posted 2010-05-26 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Epilepsy
Keywords: Epilepsy; Tracking; Electronic diary
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Epilepsy patients, electronic diary: Cohort of epilepsy patient using an electronic diary system to record all seizures, side effects, and medication compliance
  Interventions: Device: HealthBuddy
- Epilpesy patient, no electronic diary: Group of epilepsy patients who are followed using the standard of care, which is a paper diary and routine outpatient follow up visits

INTERVENTIONS:
Device: HealthBuddy — Noninvasive device for remotely reporting health information. The device does nothing to change the health of the patient, but transmits health data that is entered by the patient directly to the physician's office. Patients will enter data on seizure frequency, medication compliance, and side effects.
  Other Names: Healthbuddy is a product of Bosch Healthcare, and is already utilized in many medical institutions around the country, including the VA Health System.
  Groups: Epilepsy patients, electronic diary

SUMMARY:
The investigators propose a novel method for tracking the seizure frequency, side effect burden, and medication compliance for patients with epilepsy. The investigators intend to utilize a table-top device currently for tracking other chronic disease to collect remote data from epilepsy patients. The hypothesis is that the use of this device will lead to better longterm treatment outcomes than the standard outpatient mechanism of following patients longitudinally.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants must have a definitive diagnosis of epilepsy for at least 6 months, based on the clinical judgement of the investigators. Epilepsy is defined by two or more unprovoked seizures. Clinical history, electroencephalography, and imaging data are all instrumental in rendering a formal decision. The seizure type, frequency, or severity are not criteria for exclusion, although this information will be recorded.

Patient can range in age from birth to 65 years old; in cases of child participants, the parents are responsible for data reporting.

* Patients must have a seizure frequency of at least two seizures in a 6 month period of time.
* Patients must be on at least one anti-epileptic medication.
* Patients and/or legal guardian must be able to report seizure frequency with either a paper or electronic diary.
* Patients and/or legal guardians must be able to read and understand either English or Spanish.
* Patients and/or legal guardians must be able to complete questionnaires and provide informed consent to this study.

Exclusion Criteria:

* Exclusion criteria include: a diagnosis of psychogenic nonepileptic seizures; severe depression, anxiety, or psychosis
* Recent problem with substance abuse.

Ages: 6 Months to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be recruited from the UCSF and VAMC Outpatient Epilepsy Centers. All study participants must have a confirmed diagnosis of epilepsy (defined by two or more unprovoked seizures) for at least 6 months.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-07; Primary Completion 2011-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Seizure frequency per month | 1 year
  Assessment of seizure count accuracy by assessing total number of seizures reported per month
Medication compliance | 1 year
  Assessment of compliance with taking medications at regularly scheduled intervals
Quality of life | 1 year
  Quality of Life in Epilepsy inventory, to assess for overall change in quality of life measures

CONTACTS AND LOCATIONS:
Overall Officials: John Hixson, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Univ of California San Fran, San Francisco, California, United States